CLINICAL TRIAL: NCT02789527
Title: Exploratory Study of the Variability, in Five Human Populations, of ADME (Administration, Distribution, Metabolism, Excretion) Genotypes and Phenotypes After the Intake of the "Geneva Micrococktail"
Brief Title: Human Genomic Population Structure and Phenotype-genotype Variation in ADME Genes in Four Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Estella S. Poloni (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Estella S. Poloni, Dr, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-169
Record Dates: First submitted 2016-05-11; First posted 2016-06-03 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — Immunophenotyping; Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy volunteers in Ethiopia (Experimental): Phenotype and genotype of enzymes involved in drug metabolism in Ethiopia population
  Interventions: Drug: Phenotyping; Genetic: Genotyping
- Healthy volunteers in Oman (Experimental): Phenotype and genotype of enzymes involved in drug metabolism in Oman population
  Interventions: Drug: Phenotyping; Genetic: Genotyping
- Healthy volunteers in the Czech Republic (Experimental): Phenotype and genotype of enzymes involved in drug metabolism in Czech Republic population
  Interventions: Drug: Phenotyping; Genetic: Genotyping
- Healthy volunteers in Greece (Experimental): Phenotype and genotype of enzymes involved in drug metabolism in Greek population
  Interventions: Drug: Phenotyping; Genetic: Genotyping

INTERVENTIONS:
Drug: Phenotyping — finger-tip blood drop : enzymatic activities assessed by specific single point concentration ratios after oral intake of the Geneva micrococktail made of : CYP1A2: paraxanthine/caffeine CYP2B6: 4-hydroxybupropion/bupropion CYP2C9: 4-hydroxyflurbiprofen/flurbiprofen CYP2C19: 5-hydroxyomeprazole/omeprazole CYP2D6: dextrorphan/dextromethorphan CYP3A4: 1-hydroxymidazolam/midazolam
Genetic: Genotyping — DNA sampling from a saliva sample

SUMMARY:
Physicians know that their patients can react differently to the same medical treatment: for some of them, the drug will prove inefficient, whereas for others it might provoke side-effects, sometimes rather serious. Such differences in response to drug intake are due to several factors, of which molecular variations in specific genes, named " ADME " (Absorption, Distribution, Metabolism, Excretion). This project aims at investigating the evolutionary mechanisms responsible for the diversity of ADME genes in human populations. Because of their role at the interface between the organism and its chemical environment, ADME genes are likely targets of recent selective pressures linked to changes in the environments in which humans evolved, such as changes in dietary habits for instance.

The aim of this project is to study the diversity of ADME genes and of their expression in five populations located along a latitudinal axis that extends from East Africa to Central Europe, passing through the Arabian Peninsula and the Mediterranean area, so as to take into account environmental factors that might have influenced the evolution of this diversity. This project is thus intended to evidence the evolutionary mechanisms that shaped genomic regions that are functionally important from the clinical and epidemiological point of view. Moreover, it will allow us to extend the knowledge of human molecular diversity and its evolution to a key-region of the peopling history of our species.

ELIGIBILITY:
Inclusion Criteria:

* Women and men in good health
* Aged between 18 and 50 years
* Students or staff in the Academic Institutions where sampling will take place
* With the 2 parents and four grand-parents born to the population;
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women; or women that consider that being pregnant is a possibility;
* Allergic to one of the compounds included in micrococktail (Caffeine, Bupropion, Flurbiprofen, Omeprazole, Dextromethorphan, Midazolam, and Fexofenadine);
* Pedigree related to another volunteer participant (siblings, cousins, uncles/aunts, nephews, etc.);

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 367 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Frequencies of genotypes and haplotypes of genes involved in drug responses (240,000 Single Nucleotide Polymorphisms) in 4 human populations : 100 Ethiopian, 100 Omani, 100 Czech and 100 Greek | through study completion, an average of 2 years
  Estimation of genotype/allele/haplotype frequencies of variants in genes involved in drug responses
Activities of 6 cytochrome P450 enzymes and P-gp in 4 human populations : 100 Ethiopian, 100 Omani, 100 Czech and 100 Greek | through study completion, an average of 2 years
  Estimation of frequency distributions of classes of drug metabolizers (metabolizers' profiles: slow/normal/rapid)

SECONDARY OUTCOMES:
Comparison of frequency distributions of variants in genes involved in drug responses and of associated metabolizers' profiles in 4 human populations : 100 Ethiopian, 100 Omani, 100 Czech and 100 Greek | through study completion, an average of 3 year
  Estimation of indices of population genetic/phenotypic diversity and differentiation (expected heterozygosity, Fst). Inferences on the evolutionary mechanisms explaining the estimated diversity among and between populations.

CONTACTS AND LOCATIONS:
Overall Officials: Estella S. Poloni, Dr, Study Chair — University of Geneva/Department of Genetics and Evolution
Locations (4):
- Charles University in Prague/Faculty of Science/Department of Anthropology and Human Genetics, Prague, Czechia
- Addis Ababa University/College of Health Sciences, Addis Ababa, Ethiopia
- Democritus University of Thrace/School of Health Sciences/University Campus, Dragana, Alexandroupoli, Greece
- Sultan Qaboos University/College of Medicine and Health Sciences/Department of Pharmacology, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rollason V, Mouterde M, Daali Y, Cizkova M, Priehodova E, Kulichova I, Posova H, Petanova J, Mulugeta A, Makonnen E, Al-Habsi A, Davidson R, Al-Balushi KK, Al-Thihli K, Cerna M, Al-Yahyaee S, Cerny V, Yimer G, Poloni ES, Desmeules J. Safety of the Geneva Cocktail, a Cytochrome P450 and P-Glycoprotein Phenotyping Cocktail, in Healthy Volunteers from Three Different Geographic Origins. Drug Saf. 2020 Nov;43(11):1181-1189. doi: 10.1007/s40264-020-00983-8. PMID 32851583